CLINICAL TRIAL: NCT06253416
Title: Assessment of Muscle Thickness in Patients With Fibromyalgia and to Determine the Effectiveness of Stretching and Strengthening Exercises: a Randomized Controlled Trial
Brief Title: Assessment of Muscle Thickness in Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Pınar Özge Başaran, Principal Investigator, Hitit University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-78
Record Dates: First submitted 2024-01-24; First posted 2024-02-12 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; ultrasonography; muscle thickness; exercises
MeSH Terms: conditions — Fibromyalgia; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: prospective, randomized, single-blind, clinical study patients were randomized into two groups by a physiotherapist with sealed envelopes
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants: Patients with fibromyalgia Care provider: Physiotherapist who showed and followed the patients exercise programme Researchers were blinded to the patients groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Active Comparator): The exercise group was received a home exercise program consist of stretching and strengthening exercises, which was demonstrated by a physiotherapist and supported by visual cards. The exercises were shown to the patients in practice for at least 5 repetitions three days a week for 12 weeks. The exercise tracking form was given to the patients. The patients were called by the physiotherapist every week by telephone, and were allowed to fill out the exercise tracking form and adapt to exercise. Once every four weeks, patients were called to the hospital a total of three times and exercises were shown again in practice. Exercises started with stretching exercises; for ten seconds for three times with ten seconds of rest between each exercise. After stretching exercises extremity strengthening exercises were practiced with half-kilogram weights for the upper and lower extremities, each exercise is performed ten times with ten seconds of rest.
  Interventions: Other: Exercise
- Control group (Active Comparator): The control group was told to exercise freely and without supervision. They were advised to exercise regularly, only verbally.
  Interventions: Other: Control

INTERVENTIONS:
Other: Exercise — a home exercise program consist of stretching and strengthening exercises , 5 repetitions of each exercise three days a week for 12 weeks
  Arms: Exercise group
Other: Control — exercise freely and without supervision with their daily routine
  Arms: Control group

SUMMARY:
To investigate the muscle thickness in patients with fibromyalgia (FMS) and whether there is an increase in muscle thickness, strength, and function with stretching and strengthening exercise therapy in FMS patients.

DETAILED DESCRIPTION:
Fibromyalgia syndrome (FMS) is a common non-inflammatory disease characterized by musculoskeletal pain and is often seen in women between the ages of 40-60. Fatigue, weakness, sleep problems, depression, anxiety, and various cognitive and somatic disorders can be accompanied with widespread pain. Etiology and pathophysiology are still not clarified today. Multifactorial etiology could play a role in FMS pathogenesis. Genetic, environmental, biochemical, neuroendocrinological, psychological, muscular, peripheral/central/ autonomic nervous system, sleep disorders, immunological, and infectious factors can be suggested. Fibromyalgia is the most common rheumatological disorder after osteoarthritis in the general population and affects 2 % of the general population.

A decrease in muscle blood flow and oxygenation has been found in patients with FMS. Low levels of phosphocreatine, adenosine triphosphate and adenosine diphosphate have been observed at the sensitive point of the trapezius muscle of patients with FMS; increase in adenosine monophosphate and high creatine levels, and damage in muscle fibrils have been observed. Blood flow in muscles was measured at the time of exercise and a significant decrease was found in patients with FMS compared to healthy ones. This suggests to us that there is a relationship between symptoms and skeletal muscles in patients with FMS.

Exercise has the highest level of evidence and effective in the treatment of FMS. Most of the patients diagnosed with FMS are sedentary and their aerobic capacity is below average. According to the European League Against Rheumatism (EULAR) recommendations, exercise is definitely recommended in patients with FMS. Aerobic exercises, strengthening exercises, and stretching exercises have been shown to be beneficial. However, there is no definitive recommendation regarding the choice of exercise. The superiority of exercise types over each other is unclear. It is considered that aerobic and strengthening exercises will correct metabolic changes in muscle tissue and lead to a reduction in muscle pain, stretching and relaxation exercises reduce pain by reducing tension in soft tissues with.

The most common symptom after pain in patients with FMS is fatigue. Due to pain and fatigue, physical activity levels and muscle functions decrease. The loss of muscle function in young women is a major socioeconomic problem.

In our study, our goal is to investigate the muscle thickness and whether there is an increase in muscle thickness, muscle strength, and muscle function with stretching and strengthening exercise therapy in women with FMS.

The sample size was calculated as 30 patients for each group according to the results obtained from the power analysis (power=0.85; α=0.05; effect size= 0.70) performed with the G*Power version 3.1 program based on the values, taking into account the previous study Kapuczinski A. et al.

ELIGIBILITY:
Inclusion Criteria:

* female patients
* aged 18 to 65 years
* who were diagnosed with FMS according to the 2016 American College of Rheumatology (ACR) classification criteria

Exclusion Criteria:

* Patients who have a neurological or orthopedic disease that will prevent ambulation,
* advanced heart failure, kidney failure, liver failure, pulmonary diseases that will prevent exercise,
* inflammatory rheumatoid disease,
* pregnancy, breastfeeding, malignancy, psychiatric illness

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Muscle thickness | at the beginning of the study and again at the end of 12 weeks by the same physician.
  Muscle thickness was measured with ultrasound (6-12 Megahertz: Philips purewave, multi-frequency linear probe). The anterior thigh muscle thicknesses were evaluated on quadriceps femoris. The midpoint between the upper end of the patella and the anterior iliac anterior superior iliac spine has been determined while the patients were lying on their backs and the muscle thickness is measured from this point in centimeters. Measurements were made three times in order to avoid erroneous measurements. All measurements were performed by a single physician, who had experience in musculoskeletal US.

SECONDARY OUTCOMES:
pain level | at the beginning of the study and again at the end of 12 weeks by the same physician.
  The pain level of the patients was measured by Numerical Rating Scale (NRS). The pain in the NRS is marked on a scale such from 0 that there is no pain at all to 10 unbearable severity of pain by patients. Higher numbers indicate worst level of pain
grip strength | at the beginning of the study and again at the end of 12 weeks by the same physician.
  The grip strength was measured with a Jamar dynamo meter (Saehan hydraulic hand dynamometer). The test was performed while the patients were sitting in a chair elbow at 90 degrees of flexion and three times with each hand, with 30 seconds of rest between trials than the mean of three trials for each hand calculated separately. This instrument has a closed hydraulic system that measures the amount of grip strength produced by an isometric contraction applied to the handles and the grip strength of the hand is registered in kilograms.
Physical performance | at the beginning of the study and again at the end of 12 weeks by the same physician.
  Physical performance was assessed with the test of five times sit to stand test (FTSST) At FTSST subjects sit down without touching the back of the chair and stand up fully for 5 times as quickly as possible, and the time was measured in seconds .
Disease activity | at the beginning of the study and again at the end of 12 weeks by the same physician.
  Disease activity was evaluated with the Fibromyalgia Impact Questionnaire (FIQ). The Fibromyalgia Impact Questionnaire (FIQ) is consisting of ten items on three-factor structure with a functional, physical symptom and mental symptom domains. Each item is scored on a 11 point scale (0-10). Decreased scores indicate better disease activity. Sarmer et al. demonstrated the reliability and validity of the FIQ in the Turkish population
walking speed | at the beginning of the study and again at the end of 12 weeks by the same physician.
  walking speed was assessed with 6 meters walk test (6MWT). The 6MWT, a 6-meter flat path was marked on the hospital corridor, participants walked on the path, and walking time was measured in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: MUSTAFA KESER, Study Chair — HİTİT UNİVERSİTY EROL OLÇOK RESEARCH HOSPİTAL
Locations (1):
- Hitit University, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Due to the confidentiality of personal data